CLINICAL TRIAL: NCT03380923
Title: Precision High-Intensity Training Through Epigenetics (PHITE)
Acronym: PHITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Wright State University (Other); Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Marcas M. Bamman, PhD, Site Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: N000141613159
Record Dates: First submitted 2017-11-15; First posted 2017-12-21 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: epigenetics; exercise dose-response; inter-individual response heterogeneity; exercise training adaptations

STUDY DESIGN:
Intervention Model Description: Randomized to moderate intensity vs. high-intensity exercise training prescription.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessors analyzing biospecimen samples are blinded to the arm to which each participant has been randomly assigned when doing analysis.
  Investigators are blinded to each participant's randomized assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity (MOD) (Experimental): Endurance Training (ET): 3 d/wk x 30 minutes (min) of steady-state, moderate-intensity exercise on a treadmill or stationary cycle ergometer at target heart rate (HR) = 65-75% of maximum oxygen consumption rate (VO2max). The two modes (treadmill, bicycle) are offered for variety, and each subject is required to use each mode at least 1 d/wk to prevent bias.
  Resistance training (RT): 2 d/wk consisting of a prescription engaging all major muscle groups in 10 movements. Excluding abdominal crunches, target intensity is 12 repetitions/set to volitional fatigue. Subjects complete 3 sets of each movement, with ~60 seconds (s) rest between sets. For each movement, resistance increases when 14 repetitions are achieved for 2 of 3 sets.
  HR is monitored throughout each session and stored for analysis.
  Interventions: Behavioral: Moderate Intensity
- High Intensity (HI) (Experimental): RT: The 2 d/wk RT prescription differs from the MOD arm only in intensity and rest intervals. The same approach to progression applies, but HI RT intensity targets 8-10 repetitions per set; thus, resistance loads increase when 10 repetitions are achieved for 2 of 3 sets. The HI arm performs "superset" training, pairing movements stressing different muscle groups, with only 30-45 s between.
  ET: In lieu of steady-state endurance exercise, the HI arm performs high-intensity interval training (HIIT) 3 d/wk using a mix of challenging, explosive movements at maximal intensity. 10 x 30 s maximal intensity intervals are separated by 30 s rest intervals.
  HR is monitored throughout each session and stored for analysis.
  Interventions: Behavioral: High Intensity

INTERVENTIONS:
Behavioral: Moderate Intensity — Exercise prescription intensity is moderate
  Other Names: MOD
  Arms: Moderate Intensity (MOD)
Behavioral: High Intensity — Exercise prescription intensity is high
  Other Names: HI
  Arms: High Intensity (HI)

SUMMARY:
The PHITE collaborative team, consisting of Tim Broderick, MD (Overall PI), Wright State University (WSU); Marcas Bamman, PhD (Site PI), The University of Alabama at Birmingham (UAB); and Ron Evans, PhD and Joe Ecker, PhD, Salk Institute for Biological Studies, are working with funding from the US Department of Defense (DoD), Office of Naval Research (ONR), to explore the link between physical training and epigenetics. This is a key interest area for the DoD ONR because it provides high-impact optimization of force readiness in warfighters with diverse backgrounds.

The term epigenetics refers to heritable changes in gene expression (active versus inactive genes) that does not involve changes to the underlying DNA sequence; a change in phenotype (the set of observable characteristics of an individual resulting from the interaction of its genotype with the environment) without a change in genotype (the genetic constitution of an individual organism) . This in turn affects how cells read the genes. Epigenetic change is a regular and natural occurrence but can also be influenced by several factors including age, the environment/lifestyle, and disease state. Epigenetic modifications can manifest as commonly as the manner in which cells terminally differentiate to end up as skin cells, liver cells, brain cells, etc. New and ongoing research is continuously uncovering the role of epigenetics in a variety of human conditions. This study is designed to assess whether epigenetics is a primary mechanism modulating how individuals adapt to specific exercise training prescriptions designed to produce a warfighter phenotype.

The PHITE team is organized around a shared test population of human subjects for which UAB will oversee recruitment, training, testing, and sampling. Healthy but untrained volunteers, both men and women, 18-27 y of age-phenotypical of the US warfighter-will participate in a 12-wk, two-arm, single-blind, randomized, exercise dose-response trial comparing two intensities of combined training: Moderate-Intensity vs. High-Intensity. Biospecimens are collected before and after an acute exercise bout in the pre-training state, and again after 12 weeks of 3 d/wk combined exercise training. Numerous phenotyping assessments are collected before after the 12-week intervention period to associate exercise training outcomes with molecular changes in the skeletal muscle and blood biospecimens.

DETAILED DESCRIPTION:
Overview:

The US military relies on physical training to increase and maintain force readiness. In this study, we hypothesize that epigenetic modification is a primary mechanism by which specific physical exercise training prescriptions transduce warfighter genotype into warfighting phenotype. Our aim with this program is 3- fold. We will (1) identify training methodologies that modify epigenetic responses; (2) characterize epigenetic regulation of physiological processes, pathways and mechanisms associated with moderate and high-intensity physical training, and (3) produce real-time biomarkers of cardiorespiratory and neuromuscular performance that predict physical training outcomes. We will satisfy these goals through the following six research projects:

I. Phenotyping the Exercise Dose-Response

1. Determine the effect of exercise Intensity on neuromuscular and cardiorespiratory performance
2. Assess the impact of baseline, pre-training phenotype on acute responsiveness and adaptability to different intensity exercise regimens
3. Determine the effect of exercise intensity on mechanisms regulating muscle protein metabolism, myofiber hypertrophy, and muscle oxidative capacity

II. Real-time Genetic and Epigenetic Biomarkers of Performance

1. Identify muscle miRNA that are differentially expressed in response to varying exercise intensities
2. Identify circulating muscle-derived miRNA that are differentially expressed in response to varying exercise intensities
3. Genotype individual athletic potential for biomarker optimization

IV. Epigenomic Signatures of Human Performance

1. Identify and correlate exercise induced methylation changes in blood and muscle
2. Functionally link changes in gene expression signatures and physiologic outcomes
3. Define nuclear receptor induced epigenetic signatures in metabolically active tissues

V. Exercise Induced Histone Modifications and Chromatin Remodeling

1. Profile histone modification and histone subunit usage signatures
2. Assess chromatin as a signal integration platform for long-term stability

VI. Integrative Epigenomics

1. Categorize baseline performance and group subjects
2. Characterize epigenetic changes in response to varied exercise intensities
3. Develop forecasting models from miRNA biomarkers of performance
4. Develop epigenetic regulatory network models using Deep Belief Networks

   UAB will enroll healthy, untrained men and women who resemble the US soldier. They participate in an exercise dose response training trial that lasts approximately 12 weeks.

   There are 2 randomly assigned exercise prescriptions: MOD - 3 days per week on treadmill or stationery cycle ergometer, combined with 2 days per week of resistance training; HI - 3 days per week high intensity interval training similar to military high intensity tactical training, combined with high intensity resistance training 2 days per week.

   Physical performance is evaluated pre-training, mid-training and post-training. Additionally, body composition is evaluated pre-training and post-training. Muscle biopsies and blood draws are performed at pre-training and post-training acute exercise response bouts, and samples are sent to additional study sites for specific evaluations.

   Recruitment:

   Participants are recruited through IRB approved advertisements.

   Informed Consent:

   Once an individual is identified; meets the inclusion/exclusion criteria (pre-screen); and expresses interest in the study, a member of the research team provides the individual with a consent form to review. A member of the team follows up with the individual to further explain the study and provide an opportunity for the prospective participant to ask any questions. If the person decides to participate, he/she is scheduled for the initial visit. He/she is encouraged to ask any further questions prior to giving written informed consent.

   Participant Procedures:

   MOD exercise regimen - 3 days per week of endurance exercise at 70% heart rate reserve for 30 mins on a stationary cycle or treadmill, combined with resistance exercise on 2 of the 3 days. The resistance training prescription involves 3 sets x 10-14 repetitions for each movement, with 1 minute rest between set. The movements include leg press or squat, knee extension, chest press, overhead press, seated row, wide grip pull down, ab crunch, heel raise, triceps push down, bicep curls. Resistance loads are progressed when 14 repetitions are achieved for 2 of 3 sets. Heart rate is monitored throughout each session.

   HI Exercise regimen - 3 days per week of maximum intensity interval exercise, combined with resistance exercise on 2 of the 3 days. Instead of moderate intensity endurance exercise, participants in this group perform 10 high-intensity intervals (30 sec of work, 30 sec of rest) including box jumps, burpees, split squat jumps, kettle bell swings, cycling sprints, battle ropes, wall ball, dips, etc. The resistance training prescription involves 3 sets x 8-10 repetitions for the same movements as MOD, but with supersets of two movements. Resistance loads are progressed when 10 repetitions are achieved for 2 of 3 sets. Rest periods are 30-45 seconds between supersets. Heart rate is monitored throughout each session.

   DXA Scan -The dual energy x-ray absorptiometry (DXA) procedure for determination of body composition (muscle, fat, bone) involves minor x-ray exposure. DXA will be performed at weeks 0, and 12. The effective dose exposure is comparable to 4 hours of sun exposure

   Urine Pregnancy Test - All females who have had at least one menstrual cycle have a urine pregnancy test at initial assessment and prior to each DEXA scan. All females who have had at least one menstrual cycle are asked questions pertaining to their menstrual cycle. Because hormone levels may have significant impact on biospecimen analysis, the acute exercise bout with muscle and blood collections after the intervention period will be timed to occur in the same phase of the menstrual cycle as the pre-training acute response exercise bout.

   Muscle Sampling - A total of 7 muscle samples are collected by percutaneous needle muscle biopsy from the vastus lateralis using established procedures:

   3 collected before and after the first acute response exercise bout in the pre-training state (pre-exercise, 3 h post-exercise, 24 h post-exercise); 3 collected before and after the acute response exercise bout in the post-training state (pre-exercise, 3 h post-exercise, 24 h post-exercise);

   1 collected at a follow up visit 4 weeks after the conclusion of the intervention period.

   Blood Sampling - A total of 9 blood samples are collected by venipuncture using established procedures:

   4 collected before and after the first acute response exercise bout in the pre-training state (pre-exercise, 15 min post-exercise, 3 h post-exercise, 24 h post-exercise); 3 collected before and after the acute response exercise bout in the post-training state (pre-exercise, 15 min post-exercise, 3 h post-exercise, 24 h post-exercise);

   1 collected at a follow up visit 4 weeks after the conclusion of the intervention period.

   Exercise Performance Evaluations - 1-repetition maximum (1RM) strength on upper and lower body movements, peak aerobic capacity (VO2peak) on a cycle ergometer, Wingate anaerobic power test, peak muscle power of the knee extensors using a computer-controlled dynamometer, and vertical jump test are conducted before and after the intervention period. Some performance tests are also conducted mid-intervention (approximately week 6).

   Dietary Intake - Dietary intake will be monitored using a validated 24 hour recall at weeks 0 and 12.

   Quality Assurance:

   Exercise Sessions: Subjects will be carefully instructed in proper methods and are monitored continuously. All exercise sessions are performed under full supervision by experienced, certified staff [Certified Strength and Conditioning Specialist (National Strength and Conditioning Association) and/or Certified Exercise Specialist (American College of Sports Medicine)].

   Biospecimens Collection: All muscle biopsies and blood draws are performed by trained, professional clinician's and research staff who are experienced and locally certified.

   DXA scans: All DXA scans are performed by trained technicians at UAB.

   Genetic Testing: Genetic testing of samples will be linked to a unique participant ID that will not identify a participant in any way. Linkages to personal health information are kept secure at the clinical site (UAB).

   The research will be conducted by well trained and experienced personnel who will be identified to the IRB prior to working on this study.

   PI will be ultimately responsible for data and safety monitoring: (i) Keeping all study documents updated and available for inspection by the sponsor, UAB IRB, and other authorized reviewers; (ii) Ensuring that appropriate mechanisms to protect the safety of study participants are being followed; (iii) Ensuring adherence to protocol requirements; and (iv) Ensuring that data are accurate, complete, and secure. All documents pertaining to the conduct of the study will be kept on file by the PIs.

   Even though this trial does not meet the requirements for a Data and Safety Monitoring Board, we will follow a proactive, Data and Safety Monitoring Plan as described below.
   1. Weekly reviews at investigators/staff team meetings of recruitment progress notes, updates/reports from the exercise facility, laboratories, and data management staff, and newly available data.
   2. PIs' quarterly review of safety and interim data analysis.
   3. Annual review performed by the UAB IRB.
   4. Semi-annual patient safety review by the study team.

   All non-serious AEs will be documented, and a summary delivered to the UAB IRB at pre-determined intervals (at least annually). Any SAEs will be reported to the UAB IRB within 3 days of their discovery. Aggregate reports of AEs/SAEs will be delivered to the sponsor as mandated. If an AE (serious or non-serious) occurs, the PI will be immediately notified. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to a specialist. The study physicians will make such decisions. Depending on the type of AE/SAE, the PIs may opt to discontinue the subject from the study. The PIs will be ultimately responsible for evaluating each AE for relationship to the protocol, seriousness and expectedness, any impact on the risk-to-benefit ratio, and whether modifications are needed to the informed consent document and/or protocol. The PIs will also have the responsibility of determining whether the protocol must be suspended until satisfactory modifications are made; however, ultimate authority in such cases will rest with the UAB IRB.

ELIGIBILITY:
Inclusion Criteria:

-Healthy 18-27 year olds who are not in the US armed forces

Exclusion Criteria:

* History of regular endurance or resistance training in past 12 months
* BMI>30
* Inability to tolerate intense exercise
* Diabetes
* Uncontrolled hypertension
* Unstable or exercise induced angina pectoris or myocardial ischemia
* Vascular disease
* Neurologic disease
* Musculoskeletal disorder
* Mental health disorder
* Any chronic or infectious disease that would preclude full participation
* Lidocaine allergy
* Pregnancy

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | 16 weeks
  Muscle mass is assessed using DXA (dual-energy X-ray absorptiometry)
Change in cardiorespiratory fitness (VO2max) | 16 weeks
  VO2max is assessed using via indirect calorimetry during a graded cycle ergometry protocol

CONTACTS AND LOCATIONS:
Overall Officials: Marcas Bamman, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Center for Exercise Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available 12 months after completion of the trial. Data will be publicly available indefinitely. Data will include phenotyping test results and molecular mapping results.
Supporting Information: Study Protocol
Time Frame: De-identified data will be available 12 months after completion of the trial. Data will be publicly available indefinitely.